CLINICAL TRIAL: NCT02062385
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy, Safety, and Immunogenicity of V260 in Healthy Chinese Infants
Brief Title: Efficacy, Safety, and Immunogenicity of V260 in Healthy Chinese Infants (V260-024)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V260-024
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Rotavirus Gastroenteritis
MeSH Terms: interventions — Rotavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- V260 with staggered EPI (Experimental): V260 administered as a 2 mL oral solution at age ~2, 3, and 4 months, and staggered China Expanded Program on Immunizations (EPI) as follows: Oral poliovirus vaccine (OPV) administered as a 1 g oral solution at age ~2.5, 3.5, and 4.5 months, and diphtheria, tetanus, acellular pertussis vaccine (DTaP) administered as a 0.5 mL intramuscular injection at age ~3.5, 4.5, and 5.5 months
  Interventions: Biological: V260; Biological: OPV; Biological: DTaP
- Placebo with staggered EPI (Placebo Comparator): Placebo administered as a 2 mL oral solution at age ~2, 3, and 4 months, and staggered EPI as follows: OPV administered as a 1 g oral solution at age ~2.5, 3.5, and 4.5 months, and DTaP administered as a 0.5 mL intramuscular injection at age ~3.5, 4.5, and 5.5 months
  Interventions: Biological: Placebo to V260; Biological: OPV; Biological: DTaP
- V260 with concomitant EPI (Experimental): V260 administered as a 2 mL oral solution at age ~2, 3, and 4 months, and concomitant EPI as follows: OPV administered as a 1 g oral solution at age ~2, 3, and 4 months and DTaP administered as a 0.5 mL intramuscular injection at age ~3, 4, and 5 months
  Interventions: Biological: V260; Biological: OPV; Biological: DTaP
- Placebo with concomitant EPI (Placebo Comparator): Placebo administered as a 2 mL oral solution at age ~2, 3, and 4 months, and concomitant EPI as follows: OPV administered as a 1 g oral solution at age ~2, 3, and 4 months and DTaP administered as a 0.5 mL intramuscular injection at age ~3, 4, and 5 months
  Interventions: Biological: Placebo to V260; Biological: OPV; Biological: DTaP

INTERVENTIONS:
Biological: V260 — V260 (RotaTeq™; live, oral, pentavalent rotavirus vaccine)
  Arms: V260 with concomitant EPI; V260 with staggered EPI
Biological: Placebo to V260 — Placebo control
  Arms: Placebo with concomitant EPI; Placebo with staggered EPI
Biological: OPV — Oral poliovirus vaccine administered according to the standard of care
Biological: DTaP — Diphtheria, Tetanus, Acellular Pertussis vaccine administered according to the standard of care

SUMMARY:
This study will assess the efficacy, safety, and immunogenicity of a 3-dose regimen of RotaTeq™ (V260) in healthy Chinese infants. Approximately 4040 participants at least 6 weeks and up to 12 weeks of age at the time of the first vaccination with V260 or placebo will be enrolled and randomized (1:1) to receive either V260 or placebo. Participants will also receive the routine China Expanded Program on Immunization (EPI) vaccines (oral poliovirus vaccine [OPV] and diphtheria, tetanus, and acellular pertussis vaccine [DTaP]) either staggered or concomitantly with V260 or placebo. All participants will be followed for efficacy and safety. Immune responses to OPV and DTaP will be evaluated in a subset of participants. The primary hypothesis of the study states that V260 will be efficacious in preventing any severity of rotavirus gastroenteritis as compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants at least 6 weeks (42 days) and up to 12 weeks (84 days) of age at the time of the first study vaccination
* Parent/legal guardian agrees to participate by giving written informed consent and is willing and able to comply with study requirements

Exclusion Criteria:

* History of congenital abdominal disorders, prior rotavirus gastroenteritis, chronic diarrhea, failure to thrive, or abdominal surgery
* History of intussusception
* Impairment of immunological function, including Severe Combined Immunodeficiency (SCID)
* Acute disease, severe chronic disease, or chronic disease during the acute period
* Uncontrolled epilepsy, encephalopathy, seizure, or other progressive neurological disease
* Hypersensitivity to any component of the rotavirus vaccine, OPV, or DTaP
* Prior receipt of any rotavirus vaccine
* Fever, with an axillary temperature >=37.5 °C (or equivalent) within 24 hours before study vaccination (study vaccination can be deferred until complete resolution of febrile illness)
* Clinical evidence of active gastrointestinal illness
* Received intramuscular, oral, or intravenous corticosteroid treatment since birth (topical, ophthalmic, and inhaled steroids are permitted)
* Resides in a household with an immunocompromised person
* Receipt of a blood transfusion or blood products, including immunoglobulins
* Participation in another interventional study within 14 days before the first study vaccination or during the study
* Receipt of an investigational or non-registered product other than the study vaccine within 30 days before the first study vaccination or during the study
* For participants in immunogenicity arms: inability to obtain a blood specimen at randomization visit (note: the visit may be rescheduled so that a baseline specimen may be obtained); history of polio, diphtheria, tetanus, or pertussis disease; previous vaccination against diphtheria, tetanus, pertussis, or poliomyelitis
* Any condition which, in the opinion of the investigator, may interfere with the evaluation of the study objectives

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4040 (Actual)
Dates: Start 2014-05-30 (Actual); Primary Completion 2015-06-11 (Actual); Study Completion 2015-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mo Z, Mo Y, Li M, Tao J, Yang X, Kong J, Wei D, Fu B, Liao X, Chu J, Qiu Y, Hille DA, Nelson M, Kaplan SS. Efficacy and safety of a pentavalent live human-bovine reassortant rotavirus vaccine (RV5) in healthy Chinese infants: A randomized, double-blind, placebo-controlled trial. Vaccine. 2017 Oct 13;35(43):5897-5904. doi: 10.1016/j.vaccine.2017.08.081. Epub 2017 Sep 19. PMID 28935470
- [Derived] Mo Z, Ma X, Luo P, Mo Y, Kaplan SS, Shou Q, Zheng M, Hille DA, Arnold BA; V260-024 Study Group; Liao X. Immunogenicity of pentavalent rotavirus vaccine in Chinese infants. Vaccine. 2019 Mar 22;37(13):1836-1843. doi: 10.1016/j.vaccine.2019.02.018. Epub 2019 Feb 23. PMID 30808567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4173 participants were screened, 4040 were randomized, and 4037 received at least one dose of study vaccination.
Groups:
- V260 With Staggered EPI: V260 administered as a 2 mL oral solution at age ~2, 3, and 4 months, and staggered China Expanded Program on Immunization (EPI) as follows: Oral poliovirus vaccine (OPV) administered as a 1 g oral solution at age ~2.5, 3.5, and 4.5 months, and diphtheria, tetanus, acellular pertussis vaccine (DTaP) administered as a 0.5 mL intramuscular injection at age ~3.5, 4.5, and 5.5 months.
- V260 With Concomitant EPI: V260 administered as a 2 mL oral solution at age ~2, 3, and 4 months, and concomitant EPI as follows: OPV administered as a 1 g oral solution at age ~2, 3, and 4 months, and DTaP administered as a 0.5 mL intramuscular injection at age ~3, 4, and 5 months.
- Placebo With Concomitant EPI: Placebo administered as a 2 mL oral solution at age ~2, 3, and 4 months, and concomitant EPI as follows: OPV administered as a 1 g oral solution at age ~2, 3, and 4 months, and DTaP administered as a 0.5 mL intramuscular injection at age ~3, 4, and 5 months.
Period: Overall Study
Arm/Group | V260 With Staggered EPI | Placebo With Staggered EPI | V260 With Concomitant EPI | Placebo With Concomitant EPI
Started | 1620 | 1620 | 400 | 400
Received Vaccination 1 | 1618 | 1619 | 400 | 400
Received Vaccination 2 | 1554 | 1566 | 392 | 393
Received Vaccination 3 | 1543 | 1554 | 389 | 392
Completed | 1542 | 1555 | 388 | 391
Not Completed | 78 | 65 | 12 | 9
Not completed — Adverse Event | 19 | 13 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Incomplete EPI by database lock | 2 | 0 | 0 | 0
Not completed — Moved | 10 | 11 | 1 | 0
Not completed — Withdrawn by parent/guardian | 46 | 41 | 9 | 8
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- V260 With Staggered EPI: V260 administered as a 2 mL oral solution at age ~2, 3, and 4 months, and staggered EPI as follows: OPV administered as a 1 g oral solution at age ~2.5, 3.5, and 4.5 months, and DTaP administered as a 0.5 mL intramuscular injection at age ~3.5, 4.5, and 5.5 months.
- Total: Total of all reporting groups
Arm/Group | V260 With Staggered EPI | Placebo With Staggered EPI | V260 With Concomitant EPI | Placebo With Concomitant EPI | Total
Number analyzed (Participants) | 1620 | 1620 | 400 | 400 | 4040
Age, Continuous [Mean (Standard Deviation); unit: Days] | 57.5 (10.0) | 57.2 (9.7) | 68.3 (5.7) | 68.5 (5.7) | 59.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 806 | 775 | 185 | 183 | 1949
  Male | 814 | 845 | 215 | 217 | 2091

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Severity of Rotavirus Gastroenteritis
Description: The number of participants with rotavirus gastroenteritis (RVGE) caused by naturally-occurring wild-type rotavirus (regardless of serotype or disease severity) was assessed. The case definition of RVGE included 1) 3 or more watery or looser-than-normal stools within a 24-hour period and/or forceful vomiting, and 2) naturally-occurring wild-type rotavirus must be detected in a stool specimen taken within 7 days after the onset of symptoms.
Time Frame: From 14 days after the third dose of V260 or placebo through the first rotavirus season (up to 15 months)
Population: Participants who were vaccinated in either the staggered EPI or concomitant EPI groups, were not protocol violators, and were classified as evaluable for RVGE according to the per-protocol case definition.
Measure: Number; unit: Participants
Groups:
- V260 With Staggered or Concomitant EPI: V260 administered as a 2 mL oral solution at age ~2, 3, and 4 months, and staggered EPI as follows: OPV administered as a 1 g oral solution at age ~2.5, 3.5, and 4.5 months, and DTaP administered as a 0.5 mL intramuscular injection at age ~3.5, 4.5, and 5.5 months OR concomitant EPI as follows: OPV administered as a 1 g oral solution at age ~2, 3, and 4 months, and DTaP administered as a 0.5 mL intramuscular injection at age ~3, 4, and 5 months.
- Placebo With Staggered or Concomitant EPI: Placebo administered as a 2 mL oral solution at age ~2, 3, and 4 months, and staggered EPI as follows: OPV administered as a 1 g oral solution at age ~2.5, 3.5, and 4.5 months, and DTaP administered as a 0.5 mL intramuscular injection at age ~3.5, 4.5, and 5.5 months OR concomitant EPI as follows: OPV administered as a 1 g oral solution at age ~2, 3, and 4 months, and DTaP administered as a 0.5 mL intramuscular injection at age ~3, 4, and 5 months.
Arm/Group | V260 With Staggered or Concomitant EPI | Placebo With Staggered or Concomitant EPI
Number analyzed (Participants) | 1927 | 1937
Participants | 34 | 109
Statistical Analysis 1: Comparison: V260 With Staggered or Concomitant EPI vs Placebo With Staggered or Concomitant EPI; V260 will be considered efficacious if the lower bound of the two-sided confidence interval for efficacy is >0% at the final analysis; Test type: Superiority or Other; p < 0.001, Clopper-Pearson; To calculate the confidence interval and associated p-value, an exact conditional method based on a Poisson distribution was used; 1 - (Incidence V260 / Incidence Placebo) = 69.3, 95% CI 2-sided [54.5 to 79.7]

2. Secondary Outcome: Percentage of Participants With Elevated Temperature
Description: Elevated temperature (temperature >=37.5°C axillary or equivalent) was noted by the guardian and recorded on the Vaccination Report Card during Day 1 to Day 14 after each dose of vaccination. Elevated temperature reported by the guardian was also collected as an adverse event (pyrexia) during Day 15 to Day 30 after each dose of vaccination. The percentage of participants with axillary temperature >=37.5 °C or an adverse event of pyrexia was assessed.
Time Frame: Up to 30 days after any dose of V260 or Placebo
Population: All Subjects as Treated with follow-up specific to the endpoint
Measure: Number; unit: Percentage of participants
Arm/Group | V260 With Staggered or Concomitant EPI | Placebo With Staggered or Concomitant EPI
Number analyzed (Participants) | 2015 | 2019
Percentage of participants | 21.84 | 22.83

3. Secondary Outcome: Percentage of Participants With Vomiting or Diarrhea
Description: Episodes of vomiting and diarrhea were noted by the guardian and recorded on the Vaccination Record Card during Day 1 to Day 14 after each dose of vaccination. Vomiting and diarrhea reported by the guardian were also collected as an adverse event during Day 15 to Day 30 after any dose of vaccination. The percentage of participants with an episode or an adverse event of vomiting or diarrhea was assessed.
Time Frame: Up to 30 days after any dose of V260 or Placebo
Population: All Subjects as Treated with safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | V260 With Staggered or Concomitant EPI | Placebo With Staggered or Concomitant EPI
Number analyzed (Participants) | 2015 | 2019
Percentage of participants
  Vomiting | 2.68 | 3.52
  Diarrhea | 20.15 | 20.11

4. Secondary Outcome: Percentage of Participants With Intussusception
Description: Episodes of intussusception were collected from the time of written consent until the end of study. The percentage of participants with an episode of intussusception was assessed.
Time Frame: Up to 15 months
Population: All Subjects as Treated with safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | V260 With Staggered or Concomitant EPI | Placebo With Staggered or Concomitant EPI
Number analyzed (Participants) | 2015 | 2019
Percentage of participants | 0.10 | 0.00

5. Secondary Outcome: Number of Participants With Severe Rotavirus Gastroenteritis
Description: The number of participants with severe rotavirus gastroenteritis (RVGE) caused by naturally-occurring wild-type rotavirus (regardless of serotype or disease severity) was assessed. The case definition of RVGE included 1) 3 or more watery or looser-than-normal stools within a 24-hour period and/or forceful vomiting, and 2) naturally-occurring wild-type rotavirus must be detected in a stool specimen taken within 7 days after the onset of symptoms. Severe RVGE was defined as >=11 on the Vesikari Scoring System, a composite of the seven parameters related to symptoms and treatment with an overall range from 0 to 20.
Time Frame: From 14 days after the third dose of V260 or placebo through the first rotavirus season (up to 15 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | V260 With Staggered or Concomitant EPI | Placebo With Staggered or Concomitant EPI
Number analyzed (Participants) | 1926 | 1937
Participants | 11 | 52

6. Secondary Outcome: Percentage of Participants Who Achieved Seroprotection Against Poliovirus Type 1, 2, or 3
Description: The percentage of participants who achieved seroprotection against poliovirus Type 1, 2, or 3 was assessed. Seroprotection was defined as a neutralizing antibody titer >=1:8. This outcome was evaluated only in participants receiving concomitant administration of V260 and OPV.
Time Frame: Baseline and between 28 and 56 days after the third OPV vaccination
Population: Participants in the concomitant EPI groups who receive their scheduled doses of OPV without intervening disease specific to the antigen before the blood sample collection postdose 3, adhere to the guidelines for administration of vaccine, and have valid values available for analysis within specified day ranges.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V260 With Concomitant EPI | Placebo With Concomitant EPI
Number analyzed (Participants) | 187 | 192
Percentage of participants
  Poliovirus Type 1: Baseline, n=186, 190 | 44.09 [36.83 to 51.54] | 38.95 [31.97 to 46.27]
  Poliovirus Type 1: Post OPV #3, n=187, 192 | 98.93 [96.19 to 99.87] | 100.00 [98.10 to 100.00]
  Poliovirus Type 2: Baseline, n=186, 190 | 44.09 [36.83 to 51.54] | 41.58 [34.49 to 48.94]
  Poliovirus Type 2: Post OPV #3, n=187, 192 | 100.00 [98.05 to 100.00] | 100.00 [98.10 to 100.00]
  Poliovirus Type 3: Baseline, n=186, 190 | 25.27 [19.20 to 32.15] | 21.05 [15.49 to 27.54]
  Poliovirus Type 3: Post OPV #3, n=187, 192 | 98.93 [96.19 to 99.87] | 98.96 [96.29 to 99.87]

7. Secondary Outcome: Percentage of Participants With Any Adverse Event
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the sponsor's product, is also an adverse event.
Time Frame: Up to 30 days after any dose of V260 or Placebo
Population: All Subjects as Treated with safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | V260 With Staggered or Concomitant EPI | Placebo With Staggered or Concomitant EPI
Number analyzed (Participants) | 2015 | 2019
Percentage of participants | 53.5 | 53.3

8. Secondary Outcome: Percentage of Participants Seropositive to Diphtheria, Pertussis, or Tetanus Antigens
Description: The percentage of participants seropositive to diphtheria, pertussis, or tetanus antigens was assessed. Seropositive was defined as the following: 1) anti-diphtheria antibody titers >=0.1 International Units (IU)/mL, 2) anti-tetanus antibody titers >=0.1 IU/mL, 3) antipertussis toxin antibody titers >=20 Enzyme-linked Immunosorbent Assay (ELISA) Units (EU)/mL, 4) anti-pertussis filamentous hemagglutinin (FHA) antibody titers >=20 EU/mL. This outcome was evaluated only in participants receiving concomitant administration of V260 and EPI.
Time Frame: Baseline and between 28 and 51 days after the third DTaP vaccination
Population: Participants in the concomitant EPI groups who receive their scheduled doses of DTaP without intervening disease specific to the antigen before the blood sample collection postdose 3, adhere to the guidelines for administration of vaccine, and have valid values available for analysis within specified day ranges.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V260 With Concomitant EPI | Placebo With Concomitant EPI
Number analyzed (Participants) | 187 | 194
Percentage of participants
  Diphtheria: Baseline, n=181, 186 | 3.31 [1.23 to 7.08] | 2.69 [0.88 to 6.16]
  Diphtheria: Post DTaP #3, n=187, 194 | 99.47 [97.06 to 99.99] | 99.48 [97.16 to 99.99]
  Pertussis FHA: Baseline, n=181, 186 | 0.00 [0.00 to 2.02] | 0.00 [0.00 to 1.96]
  Pertussis FHA: Post DTaP #3, n=187, 194 | 44.92 [37.65 to 52.35] | 43.81 [36.72 to 51.10]
  Pertussis Toxin: Baseline, n=181, 186 | 1.66 [0.34 to 4.77] | 1.08 [0.13 to 3.83]
  Pertussis Toxin, Post DTaP #3, n=187, 194 | 95.19 [91.06 to 97.78] | 94.33 [90.08 to 97.14]
  Tetanus: Baseline, n=181, 186 | 12.15 [7.78 to 17.82] | 12.37 [8.00 to 17.97]
  Tetanus: Post DTaP #3, n=187, 194 | 100.00 [98.05 to 100.00] | 100.00 [98.12 to 100.00]

ADVERSE EVENTS:
Time Frame: All Adverse Events: up to 30 days after any V260 or placebo vaccination; Serious Adverse Events: from the time of written consent until the end of the study (up to 15 months)
Description: The at-risk population was All Subjects as Treated
Arm/Group | V260 With Staggered or Concomitant EPI | Placebo With Staggered or Concomitant EPI
Serious Adverse Events (participants affected / at risk) | 339/2015 | 338/2019
Other Adverse Events (participants affected / at risk) | 938/2015 | 931/2019
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V260 With Staggered or Concomitant EPI (N=2015) | Placebo With Staggered or Concomitant EPI (N=2019)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Thalassaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Thalassaemia beta (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 47 (52) | 41 (42)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 6 (6)
Intussusception (Gastrointestinal disorders) | 2 (2) | 0 (0)
Developmental delay (General disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Transient hypogammaglobulinaemia of infancy (Immune system disorders) | 2 (2) | 1 (1)
Acute tonsillitis (Infections and infestations) | 9 (9) | 5 (5)
Bronchiolitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 84 (89) | 101 (108)
Bronchopneumonia (Infections and infestations) | 129 (144) | 141 (158)
Candida infection (Infections and infestations) | 0 (0) | 3 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 20 (20) | 21 (22)
Exanthema subitum (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 7 (7) | 24 (24)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 19 (19) | 10 (10)
Herpangina (Infections and infestations) | 13 (13) | 2 (2)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Omphalitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 2 (2) | 3 (3)
Oral infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 21 (21) | 23 (23)
Pharyngitis bacterial (Infections and infestations) | 2 (2) | 5 (5)
Pneumonia (Infections and infestations) | 30 (34) | 14 (14)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 3 (3) | 3 (3)
Toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 18 (19)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rickets (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 9 (9)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V260 With Staggered or Concomitant EPI (N=2015) | Placebo With Staggered or Concomitant EPI (N=2019)
Diarrhoea (Gastrointestinal disorders) | 406 (487) | 406 (504)
Pyrexia (General disorders) | 414 (492) | 419 (481)
Nasopharyngitis (Infections and infestations) | 228 (248) | 233 (268)
Upper respiratory tract infection (Infections and infestations) | 91 (98) | 103 (114)
Cough (Respiratory, thoracic and mediastinal disorders) | 115 (133) | 92 (109)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.